CLINICAL TRIAL: NCT06290791
Title: Does a Drain Tube Influence the Postoperative Epidural Haematoma for Lumbar Biportal Endoscopic Surgery? A Randomized, Controlled Trial
Brief Title: Does a Drain Tube Influence the Postoperative Epidural Haematoma for Lumbar Biportal Endoscopic Surgery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: K2020214
Record Dates: First submitted 2024-02-27; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Drain Tube Influence the Postoperative Epidural Haematoma
Keywords: Spinal epidural hematoma; Decompression surgery; Lumbar spinal stenosis
MeSH Terms: conditions — Hematoma, Epidural, Spinal; Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (with one drain) (Experimental)
  Interventions: Procedure: two level lumbar decompression with BESS procedure received one drain.
- the group B (with two drains) (Active Comparator)
  Interventions: Procedure: two level lumbar decompression with BESS procedure received two drain.

INTERVENTIONS:
Procedure: two level lumbar decompression with BESS procedure received one drain. — patients who underwent two level lumbar decompression with BESS procedure received one drain.
  Arms: group A (with one drain)
Procedure: two level lumbar decompression with BESS procedure received two drain. — patients who underwent two level lumbar decompression with BESS procedure received two drains
  Arms: the group B (with two drains)

SUMMARY:
The purpose of this study was to evaluate if wound drains could influence postoperative spinal epidural hematoma (POSEH) in biportal endoscopic spinal surgery (BESS) procedures for decompression of lumbar spinal stenosis.

DETAILED DESCRIPTION:
How to reduce the rate of POSEH after lumbar spinal surgery is an obvious concern for spine surgeon. Wound drains were recognized as effective methods and typically used to prevent the development of symptomatic epidural hematomas after spinal surgery. However, whether range prophylactic postoperative drainage after spinal decompression for the prevention of POSEH is still controversial. Although there have been many studies focusing on the potential associations between wound drains and POSEH after lumbar spinal surgery, a prospective study focusing on the role of drains in minimally invasive surgery of BESS for lumbar spinal decompression has been rare. In present study, our team sought to investigate the influence of wound drains for POSEH and provide clinical evidence for the selection of drainage in BESS procedures for the decompression of lumbar spinal stenosis.

ELIGIBILITY:
Inclusion Criteria:

All patients with two level lumbar stenosis and neurogenic claudication with or without lumbar radiculopathy were eligible for inclusion.

Exclusion Criteria:

Patients were excluded if radiography revealed lumbar instability (motion of >3mm at the level of listhesis), if they had had previous lumbar spinal surgery, or they had American Society of Anesthesiologists (ASA) class Ⅳ or severe systemic disease.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
the cross-sectional area of POSEH | 24 hours after drain withdrawal
  the cross-sectional area of the 72th-hour POSEH after surgery

SECONDARY OUTCOMES:
the volume of drain output | 48 hours after surgery
  the total volume of the drain or drains

CONTACTS AND LOCATIONS:
Locations (1):
- Zhonglin Zhong, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhong Z, Ying J, Zhang S, Cai K, Jing X, Xu Z, Jiang L, Wu T, Wei G, Hu Q. Does the number of drain tubes influence the formation of postoperative spinal epidural hematoma following biportal endoscopic unilateral laminotomy for bilateral decompression (BE-ULBD) in patients with two-level adjacent lumbar spinal stenosis? a prospective randomized study. J Orthop Surg Res. 2025 Jun 24;20(1):615. doi: 10.1186/s13018-025-06042-1. PMID 40551242